CLINICAL TRIAL: NCT03593863
Title: The Effects of an In-school Physical Activity Intervention on Adolescents' Brain Structure and Function ('Fit to Study' Brain Imaging Sub-study)
Brief Title: The Effects of an In-school Physical Activity Intervention on Adolescents' Brain Structure and Function
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Active, not recruiting
Sponsor: University of Oxford (Other)
Collaborators: Oxford Brookes University (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Basic Science
Other Study IDs: HMR00670; EEF2681 (Other: Education Endowment Foundation)
Record Dates: First submitted 2018-05-09; First posted 2018-07-20 (Actual); Last update posted 2019-02-28 (Actual); Status verified 2018-07

CONDITIONS: Physical Activity
Keywords: Brain structure and function; Adolescents; Physical activity; Cognitive function; Mental health; Fitness
MeSH Terms: conditions — Motor Activity; Psychological Well-Being

STUDY DESIGN:
Intervention Model Description: The Fit to Study brain imaging study is embedded in the Fit to Study trial, which is a parallel group, superiority cluster-randomised efficacy trial of a 10-month (one academic year) vigorous physical activity (VPA) intervention versus control.
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- "PE as Usual" Control Group (No Intervention): The Control Group will be asked to continue with their normal PE lessons
- Intervention Group (Experimental): Physical Education (PE) Programme
  Interventions: Behavioral: Physical Education (PE) programme

INTERVENTIONS:
Behavioral: Physical Education (PE) programme — The intervention consists of a 10-month (one academic year, September-June) physical activity programme delivered by PE teachers during regular Year-8 PE lessons. The Intervention involves roughly 20 minutes of prescribed activities per week.
  Arms: Intervention Group

SUMMARY:
Physical activity has shown beneficial effects for cognitive and brain health, suggesting it may provide a highly scalable intervention to improve academic achievement. This project is part of a large-scale randomised controlled trial called Fit to Study (ClinicalTrials.gov ID: NCT03286725). The main Fit to Study trial aims to test the effect of a school-based physical activity intervention on academic performance (as well as cognition and physical measures) across Year 8 pupils in 100 secondary schools. The current study - the Fit to Study - Brain imaging sub-study - will target a sub-sample of participants in the large-scale trial, in order to test pre- to post intervention changes in hippocampal volume, as well as cognitive performance, mental health and brain organisation. We hypothesise that the intervention will change anterior hippocampal volume of Year-8 pupils, as well as mental health, cognitive performance, and more generally, brain structure and function. We further hypothesise that changes in brain organisation (e.g. hippocampal volume) may mediate changes in cognitive performance and mental health.

DETAILED DESCRIPTION:
Physical activity has shown beneficial effects for cognitive and brain health. In particular, studies have shown that physical activity has the potential to increase the volume of the anterior portion of the hippocampus, a brain structure involved in learning and memory. The Fit to Study - Brain imaging sub-study is being conducted to understand better the effects of a physical activity intervention delivered during school PE lessons on anterior hippocampal volume, as well as cognition, mental health, and brain organisation.

The Fit to Study main trial aims to test the effect of a school-based physical activity intervention on academic performance (as well as cognition and physical measures) across Year 8 pupils in 100 secondary schools. A full description of the Fit to study main trail, including its outcome measures, has been provided as part of its registration at ClinicalTrials.gov (NCT03286725).

The Fit to Study - Brain imaging sub-study will target a sub-sample of participants of the large-scale trial, in order to test pre to post intervention changes in anterior hippocampal volume, as well as cognitive performance, mental health and brain organisation. The assessments will take place pre-intervention, immediately post-intervention and 12-months post-intervention, and will comprise structural and functional magnetic resonance imaging (MRI) scans.

Fit to Study main trial participants are considered eligible for brain imaging sub-study. The brain imaging sub-study consists of two sub-samples, recruited at different times during the trial:

1. The first cohort of 60 participants completed assessments pre-intervention, will complete identical assessments post-intervention to investigate pre-to-post intervention changes, and will be invited to take part in follow-up assessments.
2. A second cohort of ~50 participants will be recruited for post-intervention assessments that are similar, but not identical, to the assessments of the first group, as well as 1-year follow-up assessments. This cohort will enable cross-sectional analysis of between-group (intervention-control) differences in a larger sample.

The assessments are similar, but not identical for the two cohorts. The key assessments are listed here and details are provided in the 'outcome measures' section.

1. Cohort 1

   * Magnetic resonance imaging (at pre- and post intervention)
   * Computer-based cognitive tasks (at pre-, and post intervention and follow-up)
   * Mental health questionnaires (at pre-, and post intervention and follow-up)
   * Physical activity assessments (at pre-, and post intervention, and follow-up)
   * Fitness assessments (at pre-, and post intervention)
   * Gait assessments (at pre- and post intervention)
2. Cohort 2

   * Magnetic resonance imaging (at post intervention only)
   * Computer-based cognitive tasks (at post intervention and follow-up)
   * Mental health questionnaires (at post intervention and follow-up)
   * Physical activity assessments (at post intervention and follow-up)
   * Gait assessments (at post-intervention only)

The primary aims of the study are:

1. To examine cross-sectional relations between anterior hippocampal volume and physical activity and fitness at baseline (cohort 1)
2. To examine whether changes in anterior hippocampal volume are greater in the intervention group compared to the control group (i.e. group by time interaction tested in cohort 1)

Secondary aims are:

1. To examine cross-sectional relations between brain structure and function, and physical activity and fitness at baseline (cohort 1)
2. To examine whether changes in brain organisation, mental health, cognitive performance and fitness are greater in the intervention group compared to the control group (i.e. group by time interaction tested in cohort 1)
3. To examine whether brain organisation, mental health, cognitive performance and fitness is different in the intervention group compared to the control group post intervention
4. To identify MRI markers predisposing the PA intervention effect

ELIGIBILITY:
1. Cohort 1:

   School level:

   Inclusion criteria
   * Enrolled in the the Fit to Study Main trial
   * Within a 75 miles radius from Oxford
   * Lower lower socio-economic background, as indicated by percentage of free school meal (FSM)-eligible pupils or postcode-derived index of multiple deprivation

   Pupil level:

   Inclusion criteria
   * Enrolled in the Fit to Study Main Trial
   * English speaking

   Exclusion criteria
   * Contraindication to MRI
   * Contraindication to VO2max fitness test
2. Cohort 2

School level:

Inclusion criteria

* High completion rates of baseline cognitive, questionnaire and fitness data relative to other schools
* Responsive to messages from the Fit to Study research team
* Lower socio-economic background, as indicated by the percentage of FSM or postcode-derived index of multiple deprivation
* For intervention schools only: adherence to the intervention.

From those schools that met criteria, a sub-sample of 10 schools is chosen by the trial manager.

Pupil level:

Inclusion criteria

* Low fitness compared to other pupils of their school who expressed an interest, based on their baseline fitness assessment (part of Fit to Study Main Trial)
* Enrolled in the Fit to Study Main Trial
* English speaking

Exclusion criteria

- Contraindication to MRI

If selected schools are not interested in the brain-imaging sub-study, these schools are replaced by other schools from the Fit to Study sample that are within reasonable travel distance (max 1.5h) from the brain imaging centre.

Ages: 11 Years to 16 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Child
Enrollment: 103 (Actual)
Dates: Start 2017-05-01 (Actual); Primary Completion 2019-09-01 (Estimated); Study Completion 2019-09-01 (Estimated)

PRIMARY OUTCOMES:
Anterior hippocampal volume (change) | 5mins, Baseline/pre-intervention (July - September 2017) and after 1 year (July - September 2018)
  Change in anterior hippocampal volume is derived using a T1-weighted magnetic resonance imaging (MRI) sequence.

SECONDARY OUTCOMES:
Structural magnetic resonance imaging | 35mins, Baseline/pre-intervention (July - September 2017) and after 1 year (May - September 2018)
  Measures of brain structure (Completed by cohort 1 and 2)
Functional magnetic resonance imaging | 15mins, Baseline/pre-intervention(July - September 2017) and after 1 year (May - September 2018)
  Measures of brain function (Completed by cohort 1 and 2)
Memory function [cognitive functioning] | 20mins, Baseline/pre-intervention (July - September 2017), after 1 year (July - September 2018) and at follow-up after 23 months (June 2018)
  Object location memory task. (This assessment is completed by cohort 1 and 2)
Memory function [cognitive functioning] | 7mins,Baseline/pre-intervention (July - September 2017), after 1 year (July - September 2018) and at follow-up after 23 months (June 2018)
  Relational memory task (This assessment is completed by cohort 1 only)
Cognitive flexibility [cognitive functioning] | 7mins, Baseline/pre-intervention (July - September 2017), after 1 year (July - September 2018) and at follow-up after 23 months (June 2018)
  Colour-shape switch task (This assessment is completed by cohort 1 only)
Planning [cognitive functioning] | 5mins, after 1 year (May-August 2018), and at follow-up after 23 months (June 2018)
  Tower of London task (This assessment is completed by cohort 2 only)
Implicit mental biases [cognitive functioning] | 20mins, Baseline/pre-intervention (July - September 2017), after 1 year (July - September 2018) and at follow-up after 23 months (June 2018)
  Mental biases are assessed using the implicit association task (This assessment is completed by cohort 1 only)
Mental health and well-being | 30mins, Baseline/pre-intervention (July - September 2017), after 1 year (July - September 2018) and at follow-up after 23 months (June 2018)
  A battery of surveys each including a number of measures:
  To assess symptoms of Attention-Deficit Hyperactivity Disorder (ADHD) a parent of the participant completed the ADHD rating scale. Puberty status is assessed using the Pubertal Development Rating Scale. Mood is assessed using the abbreviated Profile of Mood States (POMS). The abbreviated POMS scale is a questionnaire that contains 40 self-report items on a five-point Likert scale. Sleep is assessed using the Cleveland Adolescent Sleepiness Questionnaire (CASQ and the Sleep Condition Indicator (SCI). The CASQ is a self-report scale to measure excessive daytime sleepiness. The SCI is an 8-item self-report measure of insomnia symptoms.Mental health is assessed with the Strength and Difficulties Questionnaire. General health and behaviour is assessed using various items of the Health Behaviour for School Aged Children (HBSC) survey (2009/2010).
  (This battery is completed by cohort 1 and 2)
Fitness | 30mins, Baseline/pre-intervention (July - September 2017) and after 1 year (July - September 2018)
  An incremental step test on a cycle ergometer is used to measure maximal oxygen consumption (VO2max), an objective measure of cardiorespiratory fitness. (This assessment is completed by cohort 1 only)
  The 20m shuttle run (beep) test is part of the Fit to Study main trial and is therefore completed in school by both cohorts.
Objective physical activity | 7-days, Baseline/pre-intervention (September 2017), after 10 months (June/July 2018), and at follow-up after 22 months (June 2019)
  Daily average MVPA during a typical week in school term is measured using the wrist-mounted Axivity AX3 accelerometer. (This assessment is completed by cohort 1 and 2)
Gait | 5mins, Baseline/pre-intervention (July - September 2017) and after 1 year (July - September 2018)
  Participants walk over a 10m obstacle-free and flat surface walkway, while wearing a single inertial measurement unit to obtain temporal and spatial gait parameters. (This assessment is completed by cohort 1 and 2)

CONTACTS AND LOCATIONS:
Overall Officials: Heidi Johansen-Berg, Principal Investigator — University of Oxford
Locations (1):
- Wellcome Centre for Integrative Neuroimaging (WIN), Oxford, United Kingdom

IPD SHARING:
Plan to Share IPD: Undecided
The datasets generated during and/or analysed as part of the brain imaging sub-study are available from the principal investigator upon reasonable request.

REFERENCES:
- [Derived] Neil-Sztramko SE, Caldwell H, Dobbins M. School-based physical activity programs for promoting physical activity and fitness in children and adolescents aged 6 to 18. Cochrane Database Syst Rev. 2021 Sep 23;9(9):CD007651. doi: 10.1002/14651858.CD007651.pub3. PMID 34555181
- [Derived] Wassenaar TM, Wheatley CM, Beale N, Salvan P, Meaney A, Possee JB, Atherton KE, Duda JL, Dawes H, Johansen-Berg H. Effects of a programme of vigorous physical activity during secondary school physical education on academic performance, fitness, cognition, mental health and the brain of adolescents (Fit to Study): study protocol for a cluster-randomised trial. Trials. 2019 Apr 2;20(1):189. doi: 10.1186/s13063-019-3279-6. PMID 30940164